CLINICAL TRIAL: NCT05215119
Title: Comparison of Immediate with Delayed Natural Cycle Frozen Embryo Transfers from Freeze-all-IVF Cycles: a Randomized Control Trial of First Frozen Embryo Transfers
Brief Title: Immediate Versus Delayed Natural Cycle Frozen Embryo Transfers
Acronym: FET
Status: Completed | Type: Observational
Sponsor: Antalya IVF (Other)
Responsible Party: Sponsor
Other Study IDs: timetoFETJan2022
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Clinical Pregnancy
Keywords: frozen embryo transfer; time-to-transfer; natural cycle; endometrial preparation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immediate: NC endometrial preparation will start immediately after blastocyst cryopreservation confirmation.
  Interventions: Procedure: natural cycle endometrial preparation
- Delayed: NC endometrial preparation will start on day 1 of the patient's 2nd menstruation after the oocyte retrieval cycle menstruation or in a subsequent cycle.
  Interventions: Procedure: natural cycle endometrial preparation

INTERVENTIONS:
Procedure: natural cycle endometrial preparation — Cycles will be monitored from either day-10 or-12, according to patient's menstrual cycle length, with serial analysis of blood serum LH and progesterone levels and assessment of dominant follicle growth. In a spontaneous cycle, ovulation will be determined by a LH surge (>20 IU/L) and a corresponding rise in progesterone (>0.8 ng/ml). In a triggered cycle, ovulation will be determined by the administration of an hCG trigger when the dominate follicle reached >16 mm (and LH was <20 IU/L).

SUMMARY:
Introduction:

Based on recent studies the suggestion is that natural cycle frozen embryo transfers (NC FET) should preferably be used, with evidence suggesting that artificial cycle FET (AC FET) is subject to increased risks of adverse obstetric and perinatal outcomes and possibly lower live birth rates. There, however, is limited evidence on the most efficient and effective timing of NC FET following oocyte retrieval.

Objective: In this non-inferiority randomised controlled trial, the effect on reproductive outcomes of NC FET performed immediately following the oocyte retrieval cycle (i.e., after one menstruation) will be investigated.

Materials and Methods: At a single IVF centre, patients will be recruited from infertile patients presenting for freeze-all-IVF treatments. Patients aged 18 to 30 years will be enrolled, if they had ≤2 previous embryo transfers and had ≥1 blastocyst cryopreserved in their freeze-all cycles. Enrolled patients (N = 800) will be randomised (1:1) to either the immediate group (i.e., FET performed in the menstrual cycle immediately following the oocyte retrieval cycle) or the delayed group (i.e., FET performed in the menstrual cycle following two menstruations). All FET will be performed in NC. The primary outcome measure will be clinical pregnancy, defined as the visual confirmation by transvaginal ultrasound scan of a gestational sac with normal heartbeat at >5 weeks of gestation. The analyses will be performed according to per-procedure principles.

Results: The ovarian, endometrial and time to transfer outcomes of the immediate group will be compared with those of the delayed group. The clinical pregnancy rate of the immediate group will be compared with that of the delayed group.

DETAILED DESCRIPTION:
Introduction The increasing success of frozen embryo transfers (FET) in assisted reproductive technology (ART), and, therefore, the increasing use of FET to overcome standard IVF complications (i.e., adverse ovarian stimulation iatrogenesis and intra-cycle discovery of intrauterine abnormalities) and to facilitate the use of modified IVF treatment (i.e., pre-implantation genetic testing and luteal ovarian stimulation) has highlighted disadvantages inherent to FET. The major concern is the evidence that FET pregnancies are subject to adverse obstetric and perinatal outcomes such as placental and hypertensive complications, large for gestational age infants, increased pregnancy loss, increased preterm delivery. Moreover, the presumed benefits of more physiological endometria in FET demands further research into the origins of the adverse obstetric and perinatal outcomes and the elimination of their causes.

Endometrial preparation methods in FET can be divided into two major groups, artificial (AC) and natural cycle (NC) methods. While the initial studies comparing endometrial preparation methods for FET and confirmed by study reviews and meta-analyses, showed that no one method was superior in terms of reproductive outcomes, recent studies have shown that the NC cycle method results in reduced adverse obstetric and perinatal outcome rates and increased live birth rates. There is increasing evidence and understanding that using the AC method significantly increases the risks of adverse obstetric and perinatal outcomes because of the absence of a functional corpus luteum (CL). In addition to the production of hormones (i.e., estrogen and progesterone), CL also produces vasoactive molecules (i.e., relaxin, vascular endothelial growth factor) essential for optimal vascular developments in early pregnancy (i.e., implantation and placentation). Based on recent studies the suggestion, therefore, is that clinicians should preferably use NC FET. Further research, however, may be required to confirm the most optimal endometrial preparation and timing (i.e., embryo and endometrial synchrony) method for FET, because suggested preference is still being based on poor-quality evidence.

There is limited evidence on the most efficient and effective timing of NC FET following oocyte retrieval (i.e., the cycle subject to ovarian stimulation), as nearly all previous studies included the investigation of mostly AC FET. These studies, at most, confirmed that reproductive outcomes were not disadvantaged if FET were performed immediately following the oocyte retrieval cycle. Therefore, suggesting that ovarian stimulation (i.e., supraphysiological hormone levels) had no spill-over effects on endometrial and ovarian function in subsequent menstrual cycles, even in the cycle immediately following oocyte retrieval. Not having an extended delay to FET is considered by most patients to be less stressful and by clinicians to be more efficient. In this non-inferiority randomised controlled trial, the effect on reproductive outcomes of NC FET performed in menstrual cycles immediately following the oocyte retrieval cycle will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with female age 18≤40 years.
* Patients who provide written informed consent to participate in the trial and for the use of their anonymized data in research.
* Patients with <2 previous IVF treatments.
* Patients with ≥1 blastocyst cryopreserved.

Exclusion Criteria:

* Patients with female age >40 years
* Patients with female BMI ≥30 kg/m2.
* Female patients with insulin dependent diabetes or non-insulin dependent diabetes mellitus and female patients with gastrointestinal, cardiovascular, pulmonary, liver or kidney disease.
* Female patients with any contraindications or allergies to the drugs used in routine freeze-all-IVF.
* Patients with untreated intrauterine anomalies and tubal pathology.
* Patients undergoing PGT-A (aneuploidy) or PGT-M (monogenic disorders)
* Patients with no blastocysts cryopreserved.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants will be recruited from (unselected) infertile patients presenting for freeze-all-IVF treatment at the IVF centre from the start date of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy from frozen embryo transfers | Transvaginal ultrasound examination will be performed after 5 weeks of gestation (>5.5 weeks)
  Clinical pregnancy rate will be defined as a pregnancy cycle with a normal gestational sac and fetal heartbeat confirmed by ultrasound at >5.5 weeks of gestation.

SECONDARY OUTCOMES:
Pregnancy from frozen embryo transfers | Blood serum pregnancy tests will be performed 9 days after blastocyst transfer
  Pregnancy will be defined as a cycle with an arbitrary serum βHCG level of >5 mIU/mL, measured 9 days after blastocyst transfer.
Early pregnancy loss of frozen embryo transfer pregnancies | Serial transvaginal ultrasound scans will be performed to 12 weeks of gestation
  Early pregnancy loss will be defined as a pregnancy lost before 10 weeks of gestation.
Ongoing pregnancy from frozen embryo transfers | Transvaginal ultrasound scan will be performed after 12 weeks of gestation
  Ongoing pregnancy will be defined as a clinical pregnancy developing normally past 12 weeks of gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya IVF, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The
Supporting Information: Study Protocol, CSR
Time Frame: To be published immediately after publication acceptance
Access Criteria: Open access at the Mendeley Data registry at the URLs provided

REFERENCES:
- [Background] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Background] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Background] von Versen-Hoynck F, Narasimhan P, Selamet Tierney ES, Martinez N, Conrad KP, Baker VL, Winn VD. Absent or Excessive Corpus Luteum Number Is Associated With Altered Maternal Vascular Health in Early Pregnancy. Hypertension. 2019 Mar;73(3):680-690. doi: 10.1161/HYPERTENSIONAHA.118.12046. PMID 30636549
- [Background] Singh B, Reschke L, Segars J, Baker VL. Frozen-thawed embryo transfer: the potential importance of the corpus luteum in preventing obstetrical complications. Fertil Steril. 2020 Feb;113(2):252-257. doi: 10.1016/j.fertnstert.2019.12.007. PMID 32106972
- [Background] Makhijani R, Bartels C, Godiwala P, Bartolucci A, Nulsen J, Grow D, Benadiva C, Engmann L. Maternal and perinatal outcomes in programmed versus natural vitrified-warmed blastocyst transfer cycles. Reprod Biomed Online. 2020 Aug;41(2):300-308. doi: 10.1016/j.rbmo.2020.03.009. Epub 2020 Mar 21. PMID 32505542
- [Background] Pier BD, Havemann LM, Quaas AM, Heitmann RJ. Frozen-thawed embryo transfers: time to adopt a more "natural" approach? J Assist Reprod Genet. 2021 Aug;38(8):1909-1911. doi: 10.1007/s10815-021-02151-y. Epub 2021 Mar 19. PMID 33738681
- [Background] Wu H, Zhou P, Lin X, Wang S, Zhang S. Endometrial preparation for frozen-thawed embryo transfer cycles: a systematic review and network meta-analysis. J Assist Reprod Genet. 2021 Aug;38(8):1913-1926. doi: 10.1007/s10815-021-02125-0. Epub 2021 Apr 7. PMID 33829375
- [Background] Matorras R, Pijoan JI, Perez-Ruiz I, Lainz L, Malaina I, Borjaba S. Meta-analysis of the embryo freezing transfer interval. Reprod Med Biol. 2021 Jan 5;20(2):144-158. doi: 10.1002/rmb2.12363. eCollection 2021 Apr. PMID 33850447